CLINICAL TRIAL: NCT02954159
Title: Induction of Response and Remission of Vedolizumab Monotherapy Vs Combination Therapy With Tacrolimus in Patients With Moderately to Severely Active Ulcerative Colitis
Brief Title: Vedolizumab Monotherapy Vs Combination Therapy With Tacrolimus in UC
Acronym: COVET
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Andres Yarur, Assistant Professor, Dept of Gastroenterology, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-101742
Record Dates: First submitted 2016-10-14; First posted 2016-11-03 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Tacrolimus; vedolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Active Comparator): vedolizumab at standard regimen with concomitant induction treatment of tacrolimus (starting 0.05 mg per Kg twice daily)
  Interventions: Drug: Tacrolimus; Drug: Vedolizumab
- Placebo Arm (Placebo Comparator): vedolizumab at standard regimen with placebo.
  Interventions: Drug: Vedolizumab; Other: Placebo

INTERVENTIONS:
Drug: Tacrolimus — Oral tacrolimus tablet starting at 0.05mg/kg twice daily, with dose adjustments aiming for serum trough levels of 10-15 ng/ml during the first 2 weeks, and 5-10ng/ml subsequently.
  Other Names: Prograf
  Arms: Treatment arm
Drug: Vedolizumab — Intravenous Vedolizumab 300 mg at week 0, 2 and 6 followed by the same dose every 8 weeks. This drug will be given as per standard of care.
  Other Names: Entyvio
Other: Placebo — Patients will be randomized 1:1 in Treatment arm (receive Tacrolimus) and Placebo Arm.
  Arms: Placebo Arm

SUMMARY:
The aim of this study is to assess if a combination therapy of tacrolimus and vedolizumab is superior to vedolizumab monotherapy for induction of remission in moderate to severe UC, and its effect on long and short-term outcomes including colectomy rate. Secondary aim of this study is to assess the safety of tacrolimus as an induction agent in patients with UC.

DETAILED DESCRIPTION:
Phase III studies have shown that patients with UC who received vedolizumab had a higher rate of clinical response, clinical remission and mucosal healing when compared to placebo3. Nevertheless, while clinical response rate was almost 50%, the rate of clinical remission at 6 weeks was only 16.9. In comparison, in the ACT trials almost 40% of patients achieved remission at week 84. The delayed onset of action of vedolizumab monotherapy in patients with UC may lead to a higher colectomy rate and limit the use of vedolizumab in patients with active disease who require rapid induction of remission. Corticosteroids are used as a bridging agent to rapidly induce remission. However, steroid refractory or dependent disease and steroid intolerance are common. Furthermore, steroids have devastating side effects.

Tacrolimus inhibits the complexion of calcineurin with its respective cytoplasmic receptors cyclophilin and FK-binding protein 12 (FKBP-12), both of which regulate a calmodulin dependent-phosphatase. Tacrolimus has been found to be efficacious in the treatment of patients with moderate to severe UC. Unfortunately, because of the safety profile with long term use, the drug is mostly used as an induction agent.

While switching to vedolizumab from another drug that has not been efficacious or has lost effectiveness (or starting vedolizumab as a first agent) can be beneficious in the long term, patients need an induction agent in order to achieve remission in a short period of time. Tacrolimus is a widely used drug to prevent implant rejection after a transplant. Randomized controlled trials have shown that is highly effective with good response rates even after 2 weeks of therapy. In order to avoid side effects, tacrolimus is usually used for a limited amount of time (12-14 weeks), which is sufficient time to induce remission of disease. Unfortunately, as other inflammatory bowel diseases, UC recurs and patients also require a maintenance therapy. While tacrolimus has been used with good results as a long term agent, the ideal scenario is to avoid its long term use as there is still a potential for side effects and a need for a very strict close monitoring. This is why a long term maintenance agent is needed to keep the patient in remission. Until recently, no ideal agent was available for this purpose, as while anti-tumor necrosis factor agents (infliximab and adalimumab) have been approved for ulcerative colitis, its combination with another agent that induces systemic immunosuppression (in this case, tacrolimus) could potentially increase the risk of infections and/or malignancies. Because vedolizumab is gut selective, does not affect the entire immune system and post-marketing studies have confirmed its safety profile. This makes it a perfect combination agent to tacrolimus, theoretically decreasing the potential side effect while increasing its efficacy.

The hypothesis is that the addition of tacrolimus as an induction agent to a standard regimen of vedolizumab increases the efficacy of the drug, decreasing the rate of need for colectomy and other complications while quickly improving the patients' quality of life without significantly increasing the risk of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 65 years with a confirmed diagnosis of UC.
2. Diagnosis of UC established at least 6 months before enrollment or evidence of chronicity in colonic biopsies.
3. Patients with UC disease extent beyond 15 cm (must involve at least the sigmoid colon)
4. In female patients:

   * Post-menopausal for ≥1 year before screening, or
   * Surgically sterile, or
   * Agree to be on a contraceptive method from the screening visit through 4 weeks after discontinuing tacrolimus (or placebo), or
   * Completely abstain from heterosexual intercourse.
5. In male patients:

   o Agreement not to father a child through 4 weeks after discontinuing tacrolimus (through contraception or abstinence).
6. Moderate to severe UC

   * Mayo Clinic partial UC score of 6 to 12, with a baseline sigmoidoscopy sub-score of at least 2, and disease that extended 15 cm or more from the anal verge.
   * Steroid dependent patients (Appendix 1)
   * Steroid naïve or steroid responsive
7. Patients are planned to start vedolizumab as part of their clinical care.
8. 5-aminosalicilates (oral or topical) are permitted as long as the dose is stable for at least 2 weeks before screening.
9. Patients with or without previous exposure to anti-TNF agents can be included. Patients with previous exposure to anti-TNF must be off infliximab for 8 weeks and off adalimumab for 4 weeks.
10. Anti-diarrheals (eg, loperamide, diphenoxylate with atropine) for control of chronic diarrhea are not permitted.The patient must be off anti-diarrheal at the time of screening.
11. Immunosupressants (thiopurines or methotrexate) must be stopped 4 weeks prior to starting the study medications.
12. Patients with previous Clostridium Difficile infection can be included as long as they received a full course of therapy and have a negative Clostridium Difficile PCR test and are infection free for 60 days prior to screening.

Exclusion Criteria:

1. Positive stool test for parasites or stool culture for pathologic bacteria within 30 days prior to enrollment.
2. Evidence or history of Clostridium Difficile infection within 60 days prior to enrollment.
3. Active Cytomegalovirus (CMV) infection evidenced by a positive CMV PCR in serum and/or positive immunohistochemistry stain in colonic tissue.
4. Uncontrolled hypertension.
5. Chronic kidney disease (defined as a glomerular filtration rate < 60 mL/min, calculated using the Modification of Diet in Renal Disease (MDRD) formula)
6. Chronic liver disease.
7. A refractory electrolyte disorder (e.g. hypomagnesemia).
8. Persistent hypomagnesemia that does not respond to oral magnesium supplementation defined as a value <1.3 mEq/L in two separate readings, despite the administration of oral magnesium [10 meq of slow-release magnesium chloride three times per day for 48 hours].
9. Persistent hypophosphatemia defined as levels <2.2 mg/dL in two separate readings, 48 hours apart despite phosphate supplementation (sodium phosphate/potassium phosphate 500 mg up to three times daily for 48 hours).
10. Creatinine values of 1.5 mg/dL in 2 separate readings.
11. Established diagnosis of diabetes mellitus.
12. Clinical or radiological evidence of megacolon.
13. Intestinal perforation, or abdominal abscess within 3 months prior to enrollment.
14. Active clinically significant bacterial infection (within 30 days of enrollment).
15. Personal history of total or sub-total colectomy.
16. Current Pregnancy or lactation.
17. Unstable or uncontrolled medical disorder.
18. Personal history of malignant neoplasm.
19. Inability to give informed consent.
20. History of alcohol or illicit drug abuse in the previous 6 months to enrollment.
21. Patient that have received any experimental drug within 6 months prior to enrollment.
22. Patients with previous exposure to vedolizumab, cyclosporine or tacrolimus.
23. Personal history of congenital or acquired immunodeficiency (eg, common variable immunodeficiency, human immunodeficiency virus [HIV] infection, organ transplantation) excluding pharmacologic immunosuppressant.
24. Any of the following laboratory abnormalities during the screening period:

    1. Hemoglobin level <9 g/dL
    2. WBC count <3 × 109/L
    3. Lymphocyte count <0.5 × 109/L
    4. Platelet count <100 × 109/L or >1200 × 109/L
    5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 × the upper limit of normal (ULN)
25. To avoid interactions, patients on medications that induce or inhibit the Cytochrome p450 family 3, subfamily A (CYP3A) will be excluded. CYP3A inducers and inhibitors are shown in Appendix 3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andres J Yarur, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm | Placebo Arm
Started | 2 | 2
Completed | 1 | 1
Not Completed | 1 | 1
Not completed — Study ended prematurely due to low enrol | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Placebo Arm | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: Steroid-free clinical response at week 6 after starting vedolizumab, defined as a reduction in the Mayo Clinic score of at least 3 points and a decrease of at least 30% from the baseline score, with a decrease of at least 1 point on the rectal bleeding subscale or an absolute rectal bleeding score of 0 or 1 while off steroids.
Time Frame: week 6
Population: Data not collected
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Clinical Response
Description: Steroid-free clinical response at week 14 after starting vedolizumab.
Time Frame: week 14
Population: Data not collected
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Mayo UC Score
Description: total score on assessment
Time Frame: Screening, Week 2, 6, 8, 14, 30
Population: Data not collected
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Short Inflammatory Bowel Disease Questionnaire
Description: total score on assessment
Time Frame: Screening, Week 6, 14, 30
Population: Data not collected
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 20 months, 13 days
Arm/Group | Treatment Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=2) | Placebo Arm (N=2)
Increase in severity of UC symptoms (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=2) | Placebo Arm (N=2)
Intermittent tremor (Nervous system disorders) | 0 (0) | 1 (1)
clinically significant elevated creatinine (Renal and urinary disorders) | 1 (1) | 0 (0)
clinically significant low phosphorus (Endocrine disorders) | 1 (1) | 0 (0)
clinically significant low magnesium (Endocrine disorders) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Emesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
increased pain (General disorders) | 1 (1) | 0 (0)
increased diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
increase in severity of UC symptoms (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was stopped due to lack of enrollment. 4 subjects were enrolled. A Amendment was needed sooner to lessen patient burden/time or increase patient compensation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT02954159/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT02954159/Prot_SAP_002.pdf